CLINICAL TRIAL: NCT03876171
Title: Culturally Modified Family Based Therapy for Haitian Youth in South Florida
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Louis Herns Marcelin, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20180597; 1R34DA043784-01A1 (NIH)
Record Dates: First submitted 2019-03-06; First posted 2019-03-15 (Actual); Results first posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Problem Behavior
MeSH Terms: conditions — Problem Behavior

STUDY DESIGN:
Intervention Model Description: This study will develop and implement a culturally specific, family-based individual, drug use, sexual risk and delinquency risk reduction program for Haitian adolescents aged 13-17 in Miami-Dade County. The goal of the pilot study is to obtain preliminary data on CIFFTA's feasibility, cultural acceptability and efficacy.
Who Masked: Participant
Masking Description: We will test the CIFFTA model against the Standard of Care currently being offered by the Miami-Dade's Juvenile Service Department (JSD) to Haitian adolescents in their diversionary program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CIFFTA (Experimental): Family-Based Adolescent Therapy, Individual Therapy, and Psycho-educational Modules
  Interventions: Behavioral: Haitian youth family-based intervention study: family functioning; Behavioral: Haitian youth intervention study: youth psychoeducational; Behavioral: Haitian family-based intervention study: psychoeducational
- Standard of Care (Active Comparator): The Diversion Programs used by the Juvenile Services Department in Miami-Dade.
  Interventions: Behavioral: Diversion Programs

INTERVENTIONS:
Behavioral: Haitian youth family-based intervention study: family functioning — A weekly group therapy with the youth in presence of a parent or caretaker in the family.
  Arms: CIFFTA
Behavioral: Haitian youth intervention study: youth psychoeducational — Weekly one and one psychoeducational module will be delivered to the youth.
  Arms: CIFFTA
Behavioral: Haitian family-based intervention study: psychoeducational — Weekly psychoeducational module will be delivered to the adolescent to the youth in the presence of a family.
  Arms: CIFFTA
Behavioral: Diversion Programs — Youth will attend individual psychological counselling at an assigned Juvenile Services Department (JSD) diversion program.
  Arms: Standard of Care

SUMMARY:
The CIFFTA study is a unique intervention that will develop and implement a culturally-specific, family-based individual, drug use, sexual risk and delinquency risk reduction program for Haitian youth ages 13-17 in Miami-Dade County, Florida.

DETAILED DESCRIPTION:
Haitian youth in Miami-Dade County who become part of the juvenile justice system have not received culturally appropriate remediating or rehabilitative attention by that system. This study will modify a specific variety of intervention, the Culturally Informed and Flexible Family-Based Treatment for Adolescents (CIFFTA) for appropriateness in Miami's Haitian cultural contexts. This study will develop and implement a culturally specific, family-based adolescent therapy, drug use, sexual risk and delinquency risk reduction program for Haitian adolescents aged 13-17 in Miami-Dade County, Florida.

ELIGIBILITY:
Inclusion Criteria :

* Adolescents aged 13 to 17
* Place of residence is Miami-Dade
* Has Haitian ancestry
* Adolescents not incarcerated
* No prior mental health care or history of psychoactive medication
* Adolescents who have lived in the US for 3 years

Exclusion Criteria:

- Youths with a documented history of mental retardation and/or organic dysfunction.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis H Marcelin, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cela T, Marcelin LH, Waldman R, Dembo R, Demezier D, Clement R, Arcayos A, Santisteban D, Jean-Gilles M, Hogue A. Haitian and Haitian American experiences of racism and socioethnic discrimination in Miami-Dade county: At-risk and court-involved youth. Fam Process. 2023 Mar;62(1):216-229. doi: 10.1111/famp.12764. Epub 2022 Mar 10. PMID 35272392
- [Derived] Marcelin LH, Cela T, Dembo R, Jean-Gilles M, Page B, Demezier D, Clement R, Waldman R. Remote delivery of a therapeutic intervention to court-mandated youths of Haitian descent during COVID-19. J Community Psychol. 2021 Sep;49(7):2938-2958. doi: 10.1002/jcop.22559. Epub 2021 Mar 18. PMID 33734451

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment steps was as follow:
  JSD Referral=> Initial Contact (w/in 3 days of referral)=>Consent Process (w/in 7 days of referral) => Randomization (assigned condition w/in 24 hrs of consent) => Conditions 1 or 2 => Baseline Assessments (w/in 7 days of Consent).
  Condition 1: referred to Modified (at home) CIFFTA intervention group. Condition 2: referred to Standard of Care (SOC).
Pre-assignment Details: Excluded:
  Participants with prior mental health care or history of psychoactive medication Participants that are incarcerated. Participants with a documented history of mental retardation and/or organic dysfunction
Groups:
- CIFFTA: Family-Based Therapy, Individual Therapy, and Psycho-educational Modules
  Haitian youth and family-based intervention study: family functioning: A weekly group therapy with the youth, the parents and other members of the family.
  Haitian youth intervention study: youth psychoeducational: Weekly one and one psychoeducational module will be delivered to the youth.
  Haitian family intervention study: family-based psychoeducational: Weekly psychoeducational module will be delivered.
  Participants will receive the CIFFTA intervention for up to 3 months.
- Standard of Care: The Diversion Programs used by the Juvenile Services Department in Miami-Dade.
  Diversion Programs: Youth will attend individual psychological counselling at an assigned Juvenile Services Department (JSD) diversion program.
  Participants in this group will receive the standard of care for up to 3 months.
Period: Overall Study
Arm/Group | CIFFTA | Standard of Care
Started | 20 | 15
Completed | 17 | 8
Not Completed | 3 | 7
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Re-arrest | 0 | 4

BASELINE CHARACTERISTICS:
Population: Baseline data was not collected for parents/caregivers.
Groups:
- Total: Total of all reporting groups
Arm/Group | CIFFTA | Standard of Care | Total
Number analyzed (Participants) | 20 | 15 | 35
Age, Continuous [Median (Full Range); unit: years] | 15 [13 to 17] | 15 [13 to 17] | 15 [13 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 13 | 8 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African Americans | 20 | 15 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Completes the Intervention:
Description: Number of participants that complete the modules constitutes the outcome measure
Time Frame: 12 months
Population: Participants dropped out because of COVID-19 during the grant period, we could not perform some of the analyses initially proposed in the grant application. This limitation was particularly true for proposed growth curve analyses, which require larger sample sizes than the sample we ultimately recruited.
Measure: Count of Participants; unit: Participants
Arm/Group | CIFFTA | Standard of Care
Number analyzed (Participants) | 20 | 15
Participants | 17 | 8

2. Primary Outcome: Number of Participants With Sustained Abstinence in Substance Use
Description: Number of participants reporting sustained abstinence in substance use
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CIFFTA | Standard of Care
Number analyzed (Participants) | 20 | 15
Participants | 17 | 8

3. Primary Outcome: Number of Participants Who Reported Sustained Abstinence in Substance Use
Description: Participants reported sustained abstinence and assessment was done through drug test.
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CIFFTA | Standard of Care
Number analyzed (Participants) | 20 | 15
Participants | 17 | 8

4. Primary Outcome: Change in Family Functioning Assessed by the Family Environment Scale (FES)
Description: Improved connectivity and communication within the family system will be assess via a composite score using the FES questionnaire with scales ranging from 0-26 with the highest score indicating that no further intervention is needed
Time Frame: Baseline, 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CIFFTA | Standard of Care
Number analyzed (Participants) | 20 | 15
score on a scale
  Baseline | 9 (1.69) | 10 (1.54)
  12 months | 9 (1.37) | 9 (1.96)

5. Primary Outcome: Change in Conduct Disorder as Assess by Revised Behavior Problem Checklists
Description: Improvement in conduct disorder as assess in Revised Behavior Problem Checklists (RBPC) evaluating the severity of disorderly behavior with scales ranging from 0 to 2 (0=no problem; 1=mild problem; 2=severe problems)
Time Frame: baseline, 12 months
Population: The measure has 113 items and the total score ranges from 0 to 226 with higher numbers indicating more problems.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CIFFTA | Standard of Care
Number analyzed (Participants) | 20 | 15
score on a scale
  Baseline | 131 (18.48) | 128 (19.19)
  12 Months | 121 (10.30) | 124 (11.13)

6. Primary Outcome: Change in Sexual Risk Behaviors as Assess by the Comprehensive Adolescent Severity Inventory (CASI)
Description: Reduction in risky sexual activities as assess by CASI using normative data-severity scores range from 0 (never) to 3 (very often)
Time Frame: baseline, 12 months
Population: Data on risky sexual behaviors was not collected from the questionnaires. There were no participants who responded to questions relevant to this measure at both the baseline and month 12 time points, therefore change data could not be calculated.
Arm/Group | CIFFTA | Standard of Care
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Recidivism in Delinquency
Description: Number of participants that have no report of arrests from the Juvenile Services Department
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CIFFTA | Standard of Care
Number analyzed (Participants) | 20 | 15
Participants | 17 | 8

8. Secondary Outcome: Number of Participants With Peer Gang Involvement
Description: Number of participants recorded involved in peer gangs.
Time Frame: 12 months
Population: We made the strategic decision to not collect data on gang involvement because of negative sociocultural norms that prevail in the community. It was an oversight that we did not amend the protocol to reflect this decision.
Arm/Group | CIFFTA | Standard of Care
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Family Communication by Parenting Style Questionnaire (PSQ)
Description: PSQ Responses rage from 1 (never) to 6 (always)
Time Frame: baseline, 12 months
Population: Data on family communication was not collected from the questionnaires. There were no participants who responded to questions relevant to this measure at both the baseline and month 12 time points, therefore change data could not be calculated.
Arm/Group | CIFFTA | Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years
Description: Adverse events were not monitored for parents/caregivers.
Groups:
- CIFFTA: Family-Based Therapy, Individual Therapy, and Psycho-educational Modules
  Haitian youth and family-based intervention study: family functioning: A weekly group therapy with the youth, the parents and other members of the family.
  Haitian youth intervention study: youth psychoeducational: Weekly one and one psychoeducational module will be delivered to the youth.
  Haitian family intervention study: family-based psychoeducational: Weekly psychoeducational module will be delivered.
Arm/Group | CIFFTA | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/15
Other Adverse Events (participants affected / at risk) | 0/20 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/71/NCT03876171/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/71/NCT03876171/SAP_001.pdf
  • Informed Consent Form (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/71/NCT03876171/ICF_002.pdf